CLINICAL TRIAL: NCT00795353
Title: Amevive Wisdom Acquired Through Real-world Evidence - 2 (A.W.A.R.E.-2) Program: Long-Term Study
Brief Title: Assess the Long-term Effectiveness and Safety of Amevive (Alefacept) in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Acronym: AWARE-2
Status: Terminated | Type: Observational
Why Stopped: The study was terminated early due to insufficient subject enrolment in order to meet the primary and secondary endpoints
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: A.W.A.R.E.-2
Record Dates: First submitted 2008-11-11; First posted 2008-11-21 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2011-03

CONDITIONS: Chronic Plaque Psoriasis
Keywords: plaque psoriasis; psoriasis; alefacept; Amevive
MeSH Terms: conditions — Psoriasis | interventions — Alefacept

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10mL blood sample - Biomarker Substudy only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1. Amevive Exposure: Canadian subjects with moderate to severe chronic plaque psoriasis
  Interventions: Drug: Amevive exposure

INTERVENTIONS:
Drug: Amevive exposure — Commercial alefacept prescribed by Physician
  Other Names: alefacept; ASP0485

SUMMARY:
The study is a prospective, multi-centre, observational study designed to assess the long-term effectiveness and safety of alefacept in subjects with moderate to severe chronic plaque psoriasis.

DETAILED DESCRIPTION:
Study includes a bio-marker sub-study to determine differences in responders vs. non-responders. Additional consent is required for the sub-study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with moderate to severe chronic plaque psoriasis who receive a new prescription for alefacept

Exclusion Criteria:

* Subjects with a contraindication to alefacept
* Subjects with a history of cancer except for adequately treated basal cell carcinoma (maximum of 2 lesions)
* Subjects with any active cancer, including skin cancer
* Subjects having a serious local infection (eg. cellulitis, abscess) or serious systemic infection (eg. pneumonia, septicemia, tuberculosis), within the 3 months prior to the first dose of alefacept.
* Subjects known to be infected with the AIDS virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Canadian subjects with moderate to severe chronic plaque psoriasis for which Amevive is clinically indicated
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2008-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Assess the long-term effectiveness and safety of alefacept in subjects with moderate to severe chronic plaque psoriasis | 8 Weeks following last dose of each treatment course throughout study

SECONDARY OUTCOMES:
Assess the quality of life of subjects on alefacept based on completion of the Dermatology Life Quality Index | 8 Weeks following last dose of each treatment course throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Canada, Inc.
Locations (18):
- Canada (18):
  - Edmonton, Alberta
  - Winnipeg, Manitoba
  - Bathurst, New Brunswick
  - Quispamsis, New Brunswick
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - London, Ontario
  - Markham, Ontario
  - Oakville, Ontario
  - Peterborough, Ontario
  - Toronto, Ontario
  - Waterloo, Ontario
  - Welland, Ontario
  - Alma, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Saint-Hyacinthe, Quebec